CLINICAL TRIAL: NCT06910046
Title: Ground-glass Opacity-dominant Peripheral Pulmonary Lesions Diagnosis Using Confocal Laser Endomicroscopy and Shape-sensing Robotic-assisted Bronchoscopy Guided Cryobiopsy: GLASS-CLEAR Study
Brief Title: GGO-dominant PPLs Diagnosis Using CLE and ssRAB-guided Cryobiopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IS25061
Record Dates: First submitted 2025-03-26; First posted 2025-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Lung Ground-Glass Opacity
Keywords: ground-glass opacity; robotic-assisted bronchoscopy; confocal laser endomicroscopy; cryobiopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with GGO-dominant peripheral pulmonary lesions (Experimental): Approximately 119 patients with GGO-dominant PPLs who meet the inclusion and exclusion criteria will be prospectively enrolled. CLE and ssRAB-guided cryobiopsy will be performed to diagnose the lesion.
  Interventions: Diagnostic Test: CLE and ssRAB-guided cryobiopsy

INTERVENTIONS:
Diagnostic Test: CLE and ssRAB-guided cryobiopsy — All procedures are performed under general anesthesia with endotracheal intubation and mechanical ventilation. A conventional flexible bronchoscope is used to examine the subject's airway and clear the secretion. After the registration procedure is completed, the catheter of the ssRAB system is navigated to the target lesion. Cone beam computed tomography (CBCT) is used to confirm whether the target lesion has been reached. After that, an appropriate CLE probe is inserted. Right before CLE imaging, 2.5 ml of 10% fluorescein sodium is administered intravenously. CLE is then used to examine the target lesion. Based on real-time CLE imaging, the optimal biopsy location is identified and localized on the fluoroscopy. After CLE imaging, the CLE probe is retracted, followed by cryobiopsy at the same location under fluoroscopy guidance. Rapid on-site evaluation is available during the procedure to assess sample adequacy.

SUMMARY:
The purpose of the study is to evaluate the diagnostic performance and safety of cryobiopsy for ground-glass opacity (GGO)-dominant peripheral pulmonary lesions (PPLs) under the guidance of shape-sensing robotic-assisted bronchoscopy (ssRAB) combined with confocal laser endomicroscopy (CLE). Additionally, the study aims to establish CLE interpretation criteria for GGO-dominant PPLs based on histopathological characteristics and validate the proposed criteria.

DETAILED DESCRIPTION:
This is a single-arm, single-center, and prospective study. Approximately 119 patients with GGO-dominant PPLs will be enrolled to undergo CLE and ssRAB-guided cryobiopsy for the diagnosis of lesions. During the procedure, CLE will be used to examine the lesion. The primary endpoint is the diagnostic yield of the procedure. The secondary endpoints include the diagnostic accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of the procedure, CLE interpretation criteria for GGO-dominant PPLs and its diagnostic efficacy in differentiating benign from malignant lesions, and the complication rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Thin-slice chest CT showing GGO-dominant peripheral pulmonary lesions (diameter≥8mm, GGO component≥50%);
3. Suspected pulmonary malignant tumor which requires transbronchial lung biopsy for diagnosis;
4. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Diffuse GGO, suspected of benign or infectious lesions;
2. Preoperative imaging showing the target biopsy lesion adjacent to medium or large blood vessels;
3. Patients with contraindications of bronchoscopy;
4. Presence of concomitant endobronchial lesion during the bronchoscopy procedure;
5. Pregnant or lactating women;
6. Patients with known allergy for fluorescein;
7. The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 1 year
  Diagnostic yield is defined as the number of diagnostic lesions divided by the total number of lesions.

SECONDARY OUTCOMES:
Diagnostic accuracy | 1 year
  Diagnostic accuracy is calculated according to the standard definition using the classical 2*2 table.
Diagnostic sensitivity | 1 year
  Diagnostic sensitivity is calculated according to the standard definition using the classical 2*2 table. Malignancy is considered as positive.
Diagnostic specificity | 1 year
  Diagnostic specificity is calculated according to the standard definition using the classical 2*2 table. Malignancy is considered as positive.
CLE interpretation criteria for GGO-dominant PPLs and its diagnostic efficacy in differentiating benign from malignant lesions. | 1 year
  The CLE interpretation criteria for different kinds of GGO-dominant PPLs and the diagnostic accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of the proposed criteria in differentiating benign from malignant lesions.
Complication rate | 1 month
  The complications refer to the total of device or procedure related adverse events during or within 1 month after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China